CLINICAL TRIAL: NCT01624246
Title: A Phase 1, Multicenter, Open-label, Single-dose Study to Assess the Pharmacokinetics of Ceftaroline Fosamil/Avibactam in Adults With Augmented Renal Clearance
Brief Title: Pharmacokinetic Study of Ceftaroline Fosamil/Avibactam in Adults With Augmented Renal Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXL-PK-04
Record Dates: First submitted 2012-06-14; First posted 2012-06-20 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Augmented Renal Clearance (ARC); Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Ceftaroline; avibactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftaroline fosamil/Avibactam (Experimental)
  Interventions: Drug: Ceftaroline fosamil/Avibactam (CXL)

INTERVENTIONS:
Drug: Ceftaroline fosamil/Avibactam (CXL) — IV infusion of CXL (combination of ceftaroline fosamil [600 mg] plus avibactam [600 mg]) infused over 60 (± 5) minutes.

SUMMARY:
To evaluate the pharmacokinetic (PK) profiles of ceftaroline and avibactam in adults with augmented renal clearance (ARC).

DETAILED DESCRIPTION:
To evaluate the single-dose pharmacokinetic (PK) profiles of ceftaroline and avibactam following intravenous (IV) administration of ceftaroline fosamil/avibactam ("CXL") in adults with augmented renal clearance (ARC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 and ≤ 55 years old
* Augmented renal clearance, defined as:

  * Estimated CrCl ≥ 115 mL/min (calculated using modified Cockcroft-Gault, before the measured 8-hour urine collection)
  * Measured CrCl ≥ 140 mL/min (from an 8-hour urine collection)
* Hospitalized and diagnosed with SIRS, defined by at least 2 of the following:

  * Temperature (oral, rectal, tympanic, or core) > 38.5°C or < 35.0°C
  * Heart rate > 90 beats/min
  * Respiratory rate > 20 breaths/min or PaCO2 < 32 mmHg
  * Leukocytosis (> 12,000 white blood cells [WBC]/mm3), leukopenia (< 4000 WBC/mm3), or bandemia (> 10% immature neutrophils [bands] regardless of total peripheral WBC)
* Requires indwelling urinary bladder catheter per standard of care (through the end of the 8-hour urine collection)

Exclusion Criteria:

* History of any known hypersensitivity or allergic reaction to cephalosporins or any β-lactam antimicrobial (eg, penicillins)
* History of chronic kidney disease, hemodialysis, or peritoneal dialysis; or history of acute renal replacement therapy (eg, hemodialysis, hemofiltration) associated with current illness
* Suspected rhabdomyolysis or creatine kinase > 10,000 U/L
* Significant anemia defined as hemoglobin < 9 g/dL or hematocrit < 27%
* Transfusion of packed red blood cells (PRBC) or whole blood within 24 hours of study drug infusion or anticipated need for a transfusion before the last PK blood sample is collected
* If female, currently pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetic Parameters of Ceftaroline and Avibactam: Area under the plasma concentration versus time curve, Cmax, Tmax, T½, , CL, Vz, and Vss. | Up to 3 days
  The following PK parameters, if calculable, will be determined for ceftaroline, ceftaroline fosamil, ceftaroline M-1, and avibactam: area under the plasma concentration versus time curve, Cmax, time of maximum plasma drug concentration (Tmax), T½, apparent total body clearance of drug from plasma (CL), apparent volume of distribution during the terminal phase (Vz), and Vss.

SECONDARY OUTCOMES:
Safety and Tolerability of a Single Dose of IV Ceftaroline fosamil and Avibactam. | 24-36 hours after last study procedure
  Adverse events will be summarized. Vital signs (pulse, blood pressure, respiratory rate, temperature), oxygen saturation and concomitant medications will be summarized. Complete blood count (CBC) and comprehensive metabolic panel results will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Forest Laboratories
Locations (21):
- United States (19):
  - Investigational Site, Fresno, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, San Diego, California
  - Investigational Site, Stanford, California
  - Investigational Site, Hartford, Connecticut
  - Investigational Site, Washington D.C., District of Columbia
  - Investigational Site, Gainesville, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Maywood, Illinois
  - Investigational Site, Peoria, Illinois
  - Investigational Site, Duluth, Minnesota
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Neptune City, New Jersey
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Houston, Texas
- Australia (2):
  - Investigational Site, Herston, Queensland
  - Investigational Site, Southport, Queensland

REFERENCES:
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827